CLINICAL TRIAL: NCT03475784
Title: Comparison of Two Fluid Strategies for Prevention of Post-dural Puncture Headache After Cesarean Delivery
Brief Title: Two Fluid Strategies for Prevention of Post-dural Puncture Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-98-2017
Record Dates: First submitted 2018-03-17; First posted 2018-03-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted fluid therapy group (Experimental): Restrictive fluid therapy: this group will not receive fluid pre-load, and will receive intraoperative crystalloids at rate of 10 mL/Kg/hour followed by postoperative crystalloids at rate of 2mL/Kg/hour.
  Interventions: Drug: Restrictive fluid therapy
- Liberal fluid therapy group (Active Comparator): Liberal fluid therapy: this group will receive fluid pre-load (5 mL/Kg), and will receive intraoperative crystalloids at rate of 10 mL/Kg/hour followed by postoperative crystalloids at rate of 6 mL/Kg/hour.
  Interventions: Drug: Liberal fluid therapy

INTERVENTIONS:
Drug: Restrictive fluid therapy — This group will receive intraoperative crystalloids at rate of 10 mL/Kg/hour followed by postoperative crystalloids at rate of 2 mL/Kg/hour.
  Other Names: Restrictive fluids
  Arms: Restricted fluid therapy group
Drug: Liberal fluid therapy — This group will receive crystalloid preload of 5 mL/Kg, then will receive intraoperative crystalloids at rate of 10 mL/Kg/hour followed by postoperative crystalloids at rate of 6 mL/Kg/hour.
  Other Names: Liberal fluids
  Arms: Liberal fluid therapy group

SUMMARY:
Postdural puncture headache (PDPH) is a common complication after cesarean delivery (CD). The role of peri-operative fluid therapy in prophylaxis against PDPH is unclear. The aim of this work is to compare restrictive versus liberal fluid therapy in prophylaxis against PDPH after CD

DETAILED DESCRIPTION:
In this study, the investigators will compare restrictive fluid therapy and liberal fluid therapy in prophylaxis against postdural puncture headache.

The restrictive group will not receive preoperative fluid loading, and will receive intraoperative crystalloids at rate of 10 mL/Kg/hour followed by postoperative crystalloids at rate of 2 mL/Kg/hour for hours. The Liberal group will receive preoperative fluid loading of 5 mL/Kg, and will receive intraoperative crystalloids at rate of 10 mL/Kg/hour, followed by postoperative crystalloids at rate of 6 mL/Kg/hour.

Both groups will be compared regarding demographic data, total peri-operative fluids, incidence of postdural puncture headache, nausea, vomiting, and intraoperative hemodynamics (heart rate and systolic blood pressure) in addition to neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Full term
* Pregnant female
* Scheduled to elective cesarean delivery

Exclusion Criteria:

* History of migraine headache
* Hypertensive disorders of pregnancy
* Cardiac morbidities,
* Baseline systolic blood pressure < 100 mmHg
* Contraindication of regional anesthesia.
* Patients with more than one single attempt for spinal block

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Incidence of post-dural puncture headache | 48 hours
  the number of patients who develop post-dural puncture headache defined as pain scale above 4

SECONDARY OUTCOMES:
incidence of post-spinal hypotension | 60 minutes
  number of patients who develop hypotension defined as decrease of systolic blood pressure by more than 20% from the baseline reading after subarachnoid block
Wong-Baker faces pain scale | 48 hours
  Pain rating scale which is expressed by the patient starting from zero scale which corresponds to no pain, till scale 10 which corresponds to worst pain
heart rate | 24 hours
  the number of heart beats per minute
postoperative nausea and vomiting | 24 hours
  the number of patients who develop postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelbarr, Professor, Study Chair — Head of obstetric anesthesia section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No